CLINICAL TRIAL: NCT03746405
Title: Effects of Connectivity-based rTMS and State-Dependency on Amygdala Activation
Acronym: ConnecTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00101172
Record Dates: First submitted 2018-11-16; First posted 2018-11-19 (Actual); Results first posted 2020-11-05 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Amygdala Activation
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Repetitive TMS (rTMS) (Active Comparator): excitatory rTMS applied over the medial prefrontal cortex (fMRI-guided)
  Interventions: Device: repetitive transcranial magnetic stimulation
- Sham repetitive TMS (rTMS) (Sham Comparator): electrical sham coil applied over the medial prefrontal cortex (fMRI-guided)
  Interventions: Device: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — excitatory 5Hz rTMS will be used
  Arms: Repetitive TMS (rTMS)
Device: Sham repetitive transcranial magnetic stimulation — an electrical sham coil reproducing the same clicking sound and tactile sensation than the active rTMS will be used
  Arms: Sham repetitive TMS (rTMS)

SUMMARY:
Posttraumatic stress disorder (PTSD) is a highly debilitating disease with response rates to pharmacological treatment rarely exceeding 60%. Preliminary attempts have been made to use repetitive transcranial magnetic stimulation (rTMS) as a non-pharmacological treatment alternative, but thus far rTMS approaches have demonstrated only modest efficacy. A major factor contributing to these limited effects stems from the depth penetration of TMS, which is not sufficient to directly modulate deep subcortical structures, such as the amygdala, that are affected in PTSD. Moreover, while rTMS effects have been shown to be state-dependent, (i.e. vary substantially according to the neural state during stimulation), this important factor is rarely considered during the clinical application of rTMS. The current study addresses both of these limitations to improve the therapeutic efficacy of rTMS for PTSD. Here we will develop a protocol to test if connectivity-based rTMS is able to modulate amygdala activity through the functional connections with medial prefrontal cortex, taking advantage of state-dependency to enhance rTMS effects by actively engaging the amygdala through a fear perception task. BOLD activation in the amygdala and its connectivity with the frontal cortex will constitute the primary outcomes to test rTMS efficacy. Heart rate variability and skin galvanic responses, acquired during the presentation of fearful faces, will be used as continuous moderators of task engagement during rTMS. If successful, this study will pave the way for a large-scale study to investigate whether state-dependent, connectivity-based rTMS of the amygdala can improve rTMS efficacy as a clinical treatment for PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Age Restrictions: Young Group (from 18 to 35 years old)
* Use of effective method of birth control for women of childbearing capacity.
* Willing to provide informed consent.

Exclusion Criteria:

* Current or recent (within the past 6 months) history of substance abuse or dependence.
* Current serious medical illness.
* History of seizure, epilepsy, stroke, brain surgery, head injury, cranial metal implants, known structural brain lesion, devices that may be affected by rTMS or MRI (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* Inability or unwilling to give informed consent.
* Diagnosed any Axis I DSM-IV disorder (MINI, DSM-IV).
* Clinically defined neurological disorder.
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure, or currently taking medication that lowers the seizure threshold.
* Claustrophobia (MRI scanner).
* Pregnancy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-16 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lysianne Beynel, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Across the 25 enrolled participants, 7 were excluded after the first visit for different reasons such as: contraindications, too high resting motor threshold or technical difficulties
Period: Overall Study
Arm/Group | Repetitive TMS (rTMS) | Sham Repetitive TMS (rTMS)
Started (Seven subjects were excluded before the second visit (when rTMS occured) and therefore were not randomized in the active or the sham group) | 10 | 8
Completed | 7 | 6
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — technical difficulties | 0 | 2

BASELINE CHARACTERISTICS:
Population: Participants who were randomized in the active or sham group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Repetitive TMS (rTMS) | Sham Repetitive TMS (rTMS) | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: African American | 1 | 0 | 1
  Ethnicity: Asian | 5 | 3 | 8
  Ethnicity: White | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Acute Effect of a rTMS Session on Brain Activation as Measured by the Cerebral Blood Flow (Blood Oxygenation Level Dependent Signal)
Description: Blood oxygenation level dependent (BOLD) will be assessed to evaluate the acute effect of rTMS applied over the medial prefrontal cortex on the amygdala activation.
  This outcome (expressed a z-score) represents the amygdala activation, either after active rTMS or after sham rTMS.
  Higher z-scores for active than for sham rTMS indicates that amygdala activity increases after active rTMS compared to sham rTMS, on the other hand lower z-score after active rTMS vs. after Sham rTMS indicated that the amygdala activity would have been reduced with active rTMS.
Time Frame: right after the rTMS session, up to one hour
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: z score in the amygdala
Arm/Group | Repetitive TMS (rTMS) | Sham Repetitive TMS (rTMS)
Number analyzed (Participants) | 7 | 6
z score in the amygdala | 0.67 (0.48) | -0.48 (0.87)
Statistical Analysis 1: Comparison: Repetitive TMS (rTMS) vs Sham Repetitive TMS (rTMS); Hypothesis: Active rTMS applied over the node in the medial prefrontal cortex the most strongly negatively connected to the right amygdala will decrease amygdala BOLD activation compared to sham rTMS; Test type: Superiority; p = 0.03, t-test, 2 sided — Give the limited sample size, this p-value was not adjusted for multiple comparisons. The threshold for statistical significant was p < 0.05; Mean Difference (Final Values) = 1.15

ADVERSE EVENTS:
Time Frame: during rTMS application, and up to one hour after.
Arm/Group | Repetitive TMS (rTMS) | Sham Repetitive TMS (rTMS)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT03746405/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT03746405/SAP_001.pdf
  • Informed Consent Form (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT03746405/ICF_002.pdf